CLINICAL TRIAL: NCT03077750
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase II Study to Evaluate the Efficacy, Tolerability, and Safety of VBP-245 in Pediatric Subjects for the Treatment of Molluscum Contagiosum
Brief Title: A Study of VBP-245 in Pediatric Patients With Molluscum Contagiosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloce BioPharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBP-245-MCV
Record Dates: First submitted 2017-01-31; First posted 2017-03-13 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Molluscum Contagiosum
Keywords: viral skin disease
MeSH Terms: conditions — Molluscum Contagiosum; Skin Diseases, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VBP-245 (Experimental): VBP-245 Topical Gel Applied to Affected Area BID
  Interventions: Drug: VBP-245 Topical Gel
- Vehicle (Placebo Comparator): Vehicle Gel Applied to Affected Area BID
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: VBP-245 Topical Gel — Topical application BID
  Arms: VBP-245
Drug: Vehicle — Vehicle Control With No Active Pharmaceutical Ingredients
  Arms: Vehicle

SUMMARY:
A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase II Study to Evaluate the Efficacy, Tolerability, and Safety of Topical VBP-245 in Pediatric Subjects for the Treatment of Molluscum Contagiosum (VBP-245-MCV).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria:

1. Males or females aged 2-18 years at screening;
2. MC diagnosed by a general physician, dermatologist or pediatrician who refers it and treatable by a topical agent;
3. Individuals with at least 1, but not exceeding 15 molluscum selected in designated treatment area:
4. Individuals whose treatment area is located anywhere on the body except for the following prohibited areas which include: eye area (including eyelids), lips, mouth cavity, nasal cavity, inner ear, palms of the hands, soles of the feet or the anogenital area;
5. Free from any systemic or dermatologic disorder that, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse advents;
6. Free from atopic dermatitis in the treatment area that, in the opinion of the investigator, will potentially get inflamed or irritated during the course of treatment;
7. Parent or guardian able to give appropriate informed consent as determined by the approving institutional review board (IRB);
8. Individuals who are generally in good health as determined by the investigator;
9. Willingness and ability of parent or guardian to read, understand, and sign the IRB-approved informed consent form after the nature of the study has been fully explained and questions have been answered;
10. Individuals who are willing to not start any new products OTC or prescription treatments and discontinue any treatment the investigator feels may interfere with the evaluation of the test products;
11. Individuals who are willing to avoid using cosmetic products, creams, salves, or ointments to the treatment area(s);
12. Individuals who are willing and able to thoroughly follow the product use instructions, attend all the scheduled visits and successfully complete the study;
13. Individuals who are willing and able to not begin any office based treatments for the duration of the study;
14. Female subjects of childbearing age with negative pregnancy test at the enrolment time in the study;
15. Female subjects who are not breastfeeding at the enrolment time in the study;
16. Female subjects that do not intend to become pregnant during their participation in the study;
17. Female subjects with reproductive potential must agree to practice medically acceptable form of birth control during the study • Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include: o Established use of hormonal methods of contraception (oral, injected, implanted, patch or vaginal ring) Barrier methods of contraception with spermicide: condom or occlusive cap (diaphragm or cervical/Vault caps) with a spermicidal foam/gel/film/cream or suppository; o Intrauterine divide (IUD) or intrauterine system (IUS); o Surgical sterilization (vasectomy, tubal occlusion, bilateral salpingectomy); Abstinence from heterosexual intercourse; when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are NOT acceptable methods of contraception

Exclusion Criteria:

Subjects meeting the following exclusion criteria will be excluded from the study:

1. Mentally incompetent or unable or not willing to give written informed consent via parent or guardian or meet study requirements
2. Known history of hypersensitivity to topical povidone-iodine
3. Significant atopic dermatitis surrounding the molluscum contagiosum lesions as judged by the investigator
4. Individual lesions greater than 5mm in diameter
5. Pregnant, breastfeeding or unwilling to undergo an acceptable form of contraception for the duration of the study;
6. Molluscum lesions located on the eye area (including eyelids), lips, mouth cavity, nasal cavity, inner ear, palms of the hands, soles of the feet or the anogenital area;
7. Have participated in an investigational trial within 30 days prior to enrollment;
8. Have required or will require systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days prior to enrollment or during the course of the study.
9. Have any uncontrolled current infection;
10. Female subject who is pregnant, lactating planning to become pregnant, or is breastfeeding;
11. Have any chronic or acute medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk (such as an immunodeficiency or relevant genetic syndrome);
12. Have any active malignancy or are undergoing treatment for any malignancy other than non-melanoma skin cancer; Subjects viewed by the Principal Investigator as not being able to complete the study -

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Reduction in number of MCV lesions | 60 days
  Number of lesions from baseline to day 60 will be counted and the reduction in number will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Krishnan, PhD, Study Director — JSS Research
Locations (3):
- United States (3):
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Parkside Pediatrics, Greenville, South Carolina
  - Coastal Pediatrics, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No